CLINICAL TRIAL: NCT04095832
Title: The Effect of Epidural Anesthesia on the Optic Nerve Sheath Diameter in Preeclampsia: A Prospective Observational Study
Brief Title: The Effect of Epidural Anesthesia on the Optic Nerve Sheath Diameter in Preeclampsia
Acronym: ONSD
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Other Study IDs: 1908-051-1055
Record Dates: First submitted 2019-09-16; First posted 2019-09-19 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Anesthesia, Epidural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parturients with preeclampsia: Parturients who were diagnosed with preeclampsia
  Interventions: Procedure: Epidural anesthesia
- Healthy parturients: Healthy full-term parturients
  Interventions: Procedure: Epidural anesthesia

INTERVENTIONS:
Procedure: Epidural anesthesia — Epidural anesthesia using standardized technique

SUMMARY:
This study aims to assess the effect of epidural anesthesia on the optic nerve sheath diameter in parturients with preeclampsia.

DETAILED DESCRIPTION:
This prospective observational study will be performed in parturients, either with or without preeclampsia, who scheduled to undergo elective cesarean delivery under epidural anesthesia. Epidural anesthesia will be done according to the standard technique. Optic nerve sheath diameter (ONSD) will be measured before and after the epidural injection of anesthetic solutions using ultrasonography. The investigators will assess whether epidural anesthesia has effect on optic nerve sheath diameter of pregnant women, and the investigators will also compare ONSD between healthy parturients and parturients with preeclampsia. The investigators will evaluate the relationship between ONSD and disease severity of preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo planned cesarean section under epidural anesthesia if they have a singleton pregnancy, complicated by severe preeclampsia.

Severe preeclampsia was defined using the American College of Obstetricians and Gynecologist Task Force on Hypertension in Pregnancy recommendations

* Controls will be healthy pregnant women at term (>37 weeks), with a singleton pregnancy, no signs or symptoms of preeclampsia and no intrauterine fetal growth restriction, who are planned to undergo elective cesarean delivery under epidural anesthesia

Exclusion Criteria:

* Contraindication to epidural anesthesia
* Morbid cardiovascular disease
* Cerebrovascular disease
* Known fetal anomaly
* Any signs of onset of labor
* Body weight < 40 kg or body weight > 100 kg
* Height < 140cm or height > 190cm
* eye disease
* infection or trauma near the eyes
* abnormality of intracranial pressure due to Intracranial pathology

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plans to include 11 preeclamptic patients and 11 healthy pregnant women.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheath diameter (ONSD) after epidural anesthesia | 3 minutes after the completion of epidural injection of the anesthetic solutions
  measured by transocular ultrasonography

SECONDARY OUTCOMES:
Optic nerve sheath diameter (ONSD) | before epidural anesthesia, 10, 20 minutes after the completion of epidural injection of the anesthetic solutions, 10 minutes after delivery of fetus, at the end of surgery.
  measured by transocular ultrasonography
Blood pressure | on delivery day
  blood pressure in mmHg
Proteinuria | during the admission period
  The presence of Proteinuria during the admission period
Epigastric pain | during the admission period
  The occurrence of epigastric pain during the admission period
Headache | during the admission period
  The occurrence of Headache during the admission period
Visual disturbances | during the admission period
  The occurrence of Visual disturbances during the admission period
Oliguria | during the admission period
  The occurrence of Oliguria during the admission period
eclampsia | during the admission period
  The occurrence of seizure during the admission period
intracranial hemorrhage | during the admission period
  The occurrence of intracranial hemorrhage during the admission period
Serum creatinine | during the admission period
  Serum creatinine concentration
Serum albumin | during the admission period
  Serum albumin concentration
Platelet count | during the admission period
  Platelet count measured during the admission period
AST | during the admission period
  AST measured during the admission period
Apgar Score of fetus | at 1 min, 5 min
  Apgar Score of delivered fetus
Umbilical arterial pH | immediately after delivery
  pH in mmol/L, Umbilical arterial blood gas analysis
ALT | during the admission period
  ALT measured during the admission period
Umbilical arterial base excess | immediately after delivery
  base excess in mmol/L, Umbilical arterial blood gas analysis
Umbilical arterial PO2 | immediately after delivery
  PO2 in mmHg, Umbilical arterial blood gas analysis
Umbilical arterial PCO2 | immediately after delivery
  PCO2 in mmHg, Umbilical arterial blood gas analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Brzan Simenc G, Ambrozic J, Prokselj K, Tul N, Cvijic M, Mirkovic T, Lucovnik M. Ocular ultrasonography for diagnosing increased intracranial pressure in patients with severe preeclampsia. Int J Obstet Anesth. 2018 Nov;36:49-55. doi: 10.1016/j.ijoa.2018.06.005. Epub 2018 Jul 4. PMID 30057149
- [Background] Ortner CM, Krishnamoorthy V, Neethling E, Flint M, Swanevelder JL, Lombard C, Fawcus S, Dyer RA. Point-of-Care Ultrasound Abnormalities in Late-Onset Severe Preeclampsia: Prevalence and Association With Serum Albumin and Brain Natriuretic Peptide. Anesth Analg. 2019 Jun;128(6):1208-1216. doi: 10.1213/ANE.0000000000003759. PMID 31094790
- [Derived] Park SK, Kim H, Kim Y, Jang YE, Kim JT. Effect of epidural anesthesia on the optic nerve sheath diameter in patients with pre-eclampsia: a prospective observational study. Reg Anesth Pain Med. 2025 Oct 6;50(10):828-834. doi: 10.1136/rapm-2024-105444. PMID 38950931